CLINICAL TRIAL: NCT01716078
Title: The Effect of Brachial Plexus Nerve Block on Distal Peripheral Nerve Conduction
Status: Withdrawn | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Other Study IDs: 365681-8
Record Dates: First submitted 2012-10-17; First posted 2012-10-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Anesthesia
Keywords: Brachial Plexus; Nerve Block; Nerve Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the conducting ability of distal extremity nerves after a supraclavicular brachial plexus nerve block (with local anesthetic) has been placed at a more proximal location in the upper extremity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female military health care beneficiaries 18 years and older, capable of providing informed consent indicating awareness of the investigational nature of the study, in keeping with institutional policy
* Written informed consent must be obtained from each patient prior to entering the study
* Patients must be willing to have a regional anesthetic nerve block placed prior to their scheduled procedure
* Patients must be willing to have neurodiagnostic tests performed prior to placement and after placement of the regional anesthesia nerve block

Exclusion Criteria:

* Refusal to have a brachial plexus nerve block placed
* Refusal to have serial nerve conduction studies performed
* Contraindication for a regional anesthesia nerve block (allergy to local anesthetic, infection at site of injection, elevated coagulation time)
* Presence of conditions affecting the hand or arm (e.g., injury, infection) that might preclude the performance of nerve conduction studies
* Presence of known major abnormalities of nerve conduction, e.g., absent median sensory potential in a patient scheduled for carpal tunnel release
* Presence of conditions affecting the contralateral hand or arm (e.g., injury, infection) that might preclude the performance of sensory and motor studies to test block or absence of a contralateral upper extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female military health care beneficiaries age 18 years and older presenting for hand surgery and eligible for a brachial plexus nerve block will be asked to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Compund Muscle Action Potential (CMAP) amplitude | 1 day
  measured for motor studies from baseline to peak in mV

SECONDARY OUTCOMES:
Distal Latency | 1 day
  the interval between the stimulation of a compound muscle and the observed response. Normal nerve conduction velocity is above 40 m/sec in the lower extremities and above 50 m/sec in the upper extremities, but age, muscle disease, temperature, and other factors can influence the velocity.
Peak Latency | 1 day
  * This represents conduction along the majority of the axons
  * It is recorded at the peak of the waveform response
Onset Latency | 1 day
  * This represents conduction along the fastest axons
  * It is recorded at the initial deflection from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Meade, Fort Meade, Maryland, United States